CLINICAL TRIAL: NCT02682537
Title: IC-BASAROTs: Verification of a New Practice Method for More Accurate Bed-side Assessment of Individual Energy Expenditure
Brief Title: IC-BASAROTs: New Practice Method for More Accurate Bed-side Assessment of Individual Energy Expenditure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Applied Sciences Neubrandenburg (Other)
Responsible Party: Principal Investigator, Luzia Valentini, Prof. Dr., University of Applied Sciences Neubrandenburg
Other Study IDs: BB023/15
Record Dates: First submitted 2016-02-08; First posted 2016-02-15 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Healthy; Body Weight; Overweight; Thinness
Keywords: Resting energy expenditure; Calorie requirements; Indirect Calorimetry
MeSH Terms: conditions — Body Weight; Overweight; Thinness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (18):
- Female, BMI: 14,00-16,49 kg/m²: Age: 18 - 100 Years
- Female, BMI: 16,50-18,49 kg/m²: Age: 18 - 100 years
- Female, BMI: 18,50-19,99 kg/m²: Age: 18 - 100 years
- Female, BMI: 20,00-24,99 kg/m²: Age: 18 - 100 years
- Female, BMI: 25,00-29,99 kg/m²: Age: 18 - 100 years
- Female, BMI: 30,00-34,99 kg/m²: Age: 18 - 100 years
- Female, BMI: 35,00-39,99 kg/m²: Age: 18 - 100 years
- Female, BMI: 40,00-44,99 kg/m²: Age: 18 - 100 years
- Female, BMI: 45,00-49,99 kg/m²: Age: 18 - 100 years
- Male, BMI: 14,00-16,49 kg/m²: Age: 18 - 100 years
- Male, BMI: 16,50-18,49 kg/m²: Age: 18 - 100 years
- Male, BMI: 18,50-19,99 kg/m²: Age: 18 - 100 years
- Male, BMI: 20,00-24,99 kg/m²: Age: 18 - 100 years
- Male, BMI: 25,00-29,99 kg/m²: Age: 18 - 100 years
- Male, BMI: 30,00-34,99 kg/m²: Age: 18 - 100 years
- Male, BMI: 35,00-39,99 kg/m²: Age: 18 - 100 years
- Male, BMI: 40,00-44,99 kg/m²: Age: 18 - 100 years
- Male, BMI: 45,00-49,99 kg/m²: Age: 18 - 100 years

SUMMARY:
Assessment of resting energy expenditure (REE) by indirect calorimetry (IC) in 1400 healthy individuals for arithmetical transformation into an bedside tool to estimate energy requirements in dietary practice (BASAROTs). A multinational, multicenter, prospective cross-sectional study.

DETAILED DESCRIPTION:
The assessment of energy expenditure is the basic requirement for any nutritional therapy. Nevertheless, there is still no accurate, scientifically validated and practical bedside tool.

The reference method for energy expenditure measurement is indirect calorimetry (IC). High costs, time requirements and the need for trained personal are main reasons for its limited use in clinical practice. Also arithmetical calculations, such as the Harris-Benedict equation, are not widely accepted.

In general energy expenditure is often estimated by so called rules of thumbs, a method requiring only one multiplication with body weight (for example: 25 kcal/kg body weight). Sex, age and BMI are usually not considered, although they are independent predictors of energy expenditure. Thus, energy expenditure estimations are often inaccurate, especially in older and overweight/obese persons.

Therefore, it is important to develop a bedside tool that is more accurate but simple enough to be accepted by practitioners. In 2004, the Austrian Society of Clinical Nutrition published the first BMI, aged and sex adapted rule of thumbs, called BASAROTs (BMI Age Sex Adjusted Rule Of Thumbs). Those were, however, based on results of the Harris Benedict equation.

The main objective of the present study is, therefore, to replace the existing BASAROTs by BASAROTs based on actual measurements of resting energy expenditure by indirect calorimetry (IC-BASAROTs).

ELIGIBILITY:
Inclusion Criteria:

* female, male
* 18 years to 85 years
* Body Mass Index: 14,0 - 49,9 kg/m²
* Eastern Cooperative Oncology Group (ECOG) Performance Status (Grade 0 or 1)
* normal thyroid function
* subjective health in dependence of BMI (underweight, normal weight, obesity, morbid obesity)

Exclusion Criteria:

* implanted pacemaker
* amputations
* paresis (mono- and diparesis)
* Asian or African descent
* above-average physical activity (competitive sport)
* present or suspicion of malignant neoplasms (tumors, metastases, hemato-oncological diseases)
* severe diseases (organ diseases, neurological diseases)
* severe dementia (MMSE < 20 points)
* pregnancy
* participation in other trials
* subjects with expect non-compliance to protocol guidelines
* intake of:
* lithium compound
* neuroleptics: Olanzapine (Zyprexa ®), Clozapine, Sertindole, Ziprasidone, Haloperidol, Thioridazine
* anticonvulsant (Carbamazepin, Valproic Acid, Topiramate)
* noradrenalin-reuptake-inhibitor (NARI): Reboxetine , Atomoxetine
* tricyclic antidepressants (Amitryptiline, Clomipramine, Doxepin, Imipramine, Trimipramin)
* Lorcaserin
* interferon-alfa, interferon-beta
* Baclofen
* Orciprenaline
* Amiodarona
* Insulin
* corticoid therapy (oral)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Minimum sample size of n = 1400: 700 mostly healthy people (50% women, aged 18-100 years, BMI 16.5 to 39.9 kg / m²), 420 underweight individuals (50% women, 18 years to 100 years, BMI from 14.0 to 16.4 kg/m²), 280 morbidly obese (50% women,18 years to 100 years, BMI 40.0-49,9 kg/m²).
  Recruitment of volunteers is performed in the local trial centers.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
resting energy expenditure (REE) (kcal) | 15 minutes
  Assessed by indirect calorimetry

SECONDARY OUTCOMES:
blood pressure (mm Hg) | one single (baseline) measurement under standardized conditions
  upper arm measurement by certified medical device
Body temperature (°C) | one single (baseline) measurement under standardized conditions
  measured axillar, by infra-red ear thermometer and non-contact thermoscan
Heart rate (bpm) | one single (baseline) measurement under standardized conditions
  measured by heart rate band and blood pressure device
Body weight (kg) | one single (baseline) measurement under standardized conditions
  measured by electronic scale integrated in BIA device
Body height (m) | one single (baseline) measurement under standardized conditions
  measured by digital stationary stadiometer
Fat mass (FM) (kg) | one single (baseline) measurement under standardized conditions
  measured by bioelectrical impedance analysis (BIA)
Fat-free mass (FFM) (kg) | one single (baseline) measurement under standardized conditions
  measured by bioelectrical impedance Analysis (BIA)
Fat-free mass index (FFMI) (kg/m²) | one single (baseline) measurement under standardized conditions
  measured by bioelectrical impedance Analysis (BIA)
Fat mass index (FMI) (kg/m²) | one single (baseline) measurement under standardized conditions
  measured by bioelectrical impedance Analysis (BIA)
Skeletal muscle mass (SMM) (kg) | one single (baseline) measurement under standardized conditions
  measured by bioelectrical impedance Analysis (BIA)
Total body water (TBW) (l) | one single (baseline) measurement under standardized conditions
  measured by bioelectrical impedance Analysis (BIA)
Extracellular water (ECW) (l) | one single (baseline) measurement under standardized conditions
  measured by bioelectrical impedance Analysis (BIA)
Resistance (R) (Ω) | one single (baseline) measurement under standardized conditions
  measured by bioelectrical impedance Analysis (BIA)
Reactance (Xc) (Ω) | one single (baseline) measurement under standardized conditions
  measured by bioelectrical impedance Analysis (BIA)
Phase angle (°) | one single (baseline) measurement under standardized conditions
  measured by bioelectrical impedance Analysis (BIA)
Waist circumference (cm) | one single (baseline) measurement under standardized conditions
  measured by measuring tape
International Physical Activity Questionnaire (IPAQ) short form | one single (baseline) interview

CONTACTS AND LOCATIONS:
Overall Officials: Luzia Valentini, Prof. Dr., Principal Investigator — Neubrandenburg University of Applied Sciences
Locations (6):
- Germany (6):
  - Technical University of Munich, Munich, Bavaria
  - Fulda University of Applied Sciences, Fulda, Hesse
  - Dietrich Bonheoffer Hospital of Neubrandenburg, Neubrandenburg, Mecklenburg-Vorpommern
  - University of Applied Sciences Neubrandenburg, Neubrandenburg, Mecklenburg-Vorpommern
  - Profil Institut for Metabolic Research, Mainz, Rhineland-Palatinate
  - Leipzig University - Medical Center IFB AdiposityDiseases, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: Yes
The other study centers forward us pseudonymised participant data for evaluation. It might also be possible that we share selected pseudonymised participant data with the other study centers.

REFERENCES:
- [Background] Elizabeth Weekes C. Controversies in the determination of energy requirements. Proc Nutr Soc. 2007 Aug;66(3):367-77. doi: 10.1017/S0029665107005630. PMID 17637089
- [Background] Schoeller DA. Making indirect calorimetry a gold standard for predicting energy requirements for institutionalized patients. J Am Diet Assoc. 2007 Mar;107(3):390-2. doi: 10.1016/j.jada.2007.01.030. No abstract available. PMID 17324655
- [Background] Valentini L, Roth E, Jadrna K, Postrach E, Schulzke JD. The BASA-ROT table: an arithmetic-hypothetical concept for easy BMI-, age-, and sex-adjusted bedside estimation of energy expenditure. Nutrition. 2012 Jul;28(7-8):773-8. doi: 10.1016/j.nut.2011.11.020. PMID 22704700
- [Background] Lawrence M. Predicting energy requirements: is energy expenditure proportional to the BMR or to body weight? An analysis of data collected in rural Gambian women. Eur J Clin Nutr. 1988 Nov;42(11):919-27. PMID 3074920
- [Background] Piers LS, Soares MJ, McCormack LM, O'Dea K. Is there evidence for an age-related reduction in metabolic rate? J Appl Physiol (1985). 1998 Dec;85(6):2196-204. doi: 10.1152/jappl.1998.85.6.2196. PMID 9843543
- [Background] Muller MJ, Bosy-Westphal A, Kutzner D, Heller M. Metabolically active components of fat-free mass and resting energy expenditure in humans: recent lessons from imaging technologies. Obes Rev. 2002 May;3(2):113-22. doi: 10.1046/j.1467-789x.2002.00057.x. PMID 12120418
- [Background] Dickerson RN. Optimal caloric intake for critically ill patients: first, do no harm. Nutr Clin Pract. 2011 Feb;26(1):48-54. doi: 10.1177/0884533610393254. PMID 21266697
- [Background] Berger MM, Pichard C. Development and current use of parenteral nutrition in critical care - an opinion paper. Crit Care. 2014 Aug 8;18(4):478. doi: 10.1186/s13054-014-0478-0. PMID 25184816
- [Background] Heidegger CP, Berger MM, Graf S, Zingg W, Darmon P, Costanza MC, Thibault R, Pichard C. Optimisation of energy provision with supplemental parenteral nutrition in critically ill patients: a randomised controlled clinical trial. Lancet. 2013 Feb 2;381(9864):385-93. doi: 10.1016/S0140-6736(12)61351-8. Epub 2012 Dec 3. PMID 23218813
- [Background] Bader N, Bosy-Westphal A, Dilba B, Muller MJ. Intra- and interindividual variability of resting energy expenditure in healthy male subjects -- biological and methodological variability of resting energy expenditure. Br J Nutr. 2005 Nov;94(5):843-9. doi: 10.1079/bjn20051551. PMID 16277790
- [Background] Bosy-Westphal A, Eichhorn C, Kutzner D, Illner K, Heller M, Muller MJ. The age-related decline in resting energy expenditure in humans is due to the loss of fat-free mass and to alterations in its metabolically active components. J Nutr. 2003 Jul;133(7):2356-62. doi: 10.1093/jn/133.7.2356. PMID 12840206
- [Background] Gonnissen HK, Adam TC, Hursel R, Rutters F, Verhoef SP, Westerterp-Plantenga MS. Sleep duration, sleep quality and body weight: parallel developments. Physiol Behav. 2013 Sep 10;121:112-6. doi: 10.1016/j.physbeh.2013.04.007. Epub 2013 May 3. PMID 23643826
- [Background] Chaput JP, St-Onge MP. Increased food intake by insufficient sleep in humans: are we jumping the gun on the hormonal explanation? Front Endocrinol (Lausanne). 2014 Jul 15;5:116. doi: 10.3389/fendo.2014.00116. eCollection 2014. No abstract available. PMID 25076940
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Rutten A, Abu-Omar K. Prevalence of physical activity in the European Union. Soz Praventivmed. 2004;49(4):281-9. doi: 10.1007/s00038-004-3100-4. PMID 15357531
- [Background] Bosy-Westphal A, Schautz B, Later W, Kehayias JJ, Gallagher D, Muller MJ. What makes a BIA equation unique? Validity of eight-electrode multifrequency BIA to estimate body composition in a healthy adult population. Eur J Clin Nutr. 2013 Jan;67 Suppl 1:S14-21. doi: 10.1038/ejcn.2012.160. PMID 23299866